CLINICAL TRIAL: NCT02656758
Title: A Randomized Controlled Study on the Effect of Intensive Functional Training on Children With Attention Deficit Hyperactivity Disorder
Brief Title: Intensive Executive Function Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ZIli Fan (Other)
Responsible Party: Sponsor-Investigator, ZIli Fan, postgraduate, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z151100004015103
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Executive function training (Experimental): the experimental group will receive 12 sessions of intensive Executive function training weekly immediately
  Interventions: Behavioral: intensive Executive function training
- the waitlist group (Other): the waitlist group will wait 12 weeks before receiving intensive executive function training for comparison.
  Interventions: Behavioral: intensive Executive function training

INTERVENTIONS:
Behavioral: intensive Executive function training — Children diagnosis of attention deficit hyperactivity disorder are randomized to the experimental condition(Executive Function training) or waiting group experimental:participants will receive 12 sessions of intensive executive function training weekly no intervention :waiting participants will not be treated with intensive executive function training and keep waiting for 12 weeks for comparison

SUMMARY:
The investigators intent to recruit 80 attention deficit hyperactivity disorder families. The attention deficit hyperactivity disorder families had received executive function training one year before.They will be randomized to intervention group and control group using a block randomization design. The intervention group will participate in intensive executive function training immediately,while the control group will receive executive training after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of child attention deficit hyperactivity disorder
* full-scale intelligence quotient (FSIQ) ≥70
* stable on medication for attention deficit hyperactivity disorder children at least 3 months
* participation in the early implementation of functional training one year before

Exclusion Criteria:

* individuals with major neurological disorders
* a diagnosis of schizophrenia, epilepsy, mental retardation or other brain disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in attention deficit hyperactivity disorder-rating scale | baseline, after the training (12 weeks)

SECONDARY OUTCOMES:
Change in behavior rating scale of executive function | baseline, after the training (12 weeks)
Cambridge Neuropsychological Test Automatic Battery | baseline, after the training (12 weeks)
Behavior Rating Inventory of Executive Function | baseline, after the training (12week)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Qian, Principal Investigator — Peking University Sixth Hospital/Institute of Mental Health
Locations (1):
- Peking University Sixth Hospital/Institute of Mental Health, Beijing, Beijing Municipality, China